CLINICAL TRIAL: NCT04294537
Title: TAP Block or Wound Infiltration for Laparoscopic Pediatric Appendectomy: Prospective Randomized Study
Brief Title: TAP Block or Wound Infiltration for Laparoscopic Pediatric Appendectomy: a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ospedale di Circolo - Fondazione Macchi (Other)
Responsible Party: Principal Investigator, Andrea Luigi Ambrosoli, Anesthesia and Intensive Care Chief - Ospedale Filippo Del Ponte, Ospedale di Circolo - Fondazione Macchi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VARPON001
Record Dates: First submitted 2019-11-09; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Appendectomy; Laparoscopy; Anesthesia, Conduction; Child, Preschool
Keywords: TAP Block; Wound Infiltration; Laparoscopic Appendectomy; Levobupivacaine; Pediatric Surgery; Pediatric Anesthesia
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block (Experimental): Bilateral ultrasound-guided single-shot TAP block with 0,15% levobupivacaine 0,75 mg/kg per side.
  Interventions: Procedure: TAP Block; Procedure: General anesthesia; Drug: Postperative analgesia
- LIA - local wound infiltration (Active Comparator): Wound infiltration with 0,5% levobupivacaine 1.5 mg/kg
  Interventions: Procedure: LIA local infiltration; Procedure: General anesthesia; Drug: Postperative analgesia

INTERVENTIONS:
Procedure: TAP Block — At the end of surgery patients will receive bilateral ultrasound-guided single-shot TAP block: 0,15% levobupivacaine 0,75 mg/kg per side will be injected between internal oblique and transveralis fascia
  Arms: TAP block
Procedure: LIA local infiltration — At the end of surgery 0,5% levobupivacaine 1.5 mg/kg, equally distributed between ports, injected in the skin and subcutaneous tissue during wound closure.
  Arms: LIA - local wound infiltration
Procedure: General anesthesia — General anesthesia will be induced with fentanyl 1,5 mcg/kg, propofol 2 mg/kg, rocuronium 0,6 mg/kg; after intubation anesthesia will be mantained with sevoflurane (MAC 1).
  30 minutes after induction will be administered paracetamol 15 mg/kg iv.
Drug: Postperative analgesia — During first 48 hours after surgery all patients wil receive paracetamol 15 mg/kg iv every 8 hours and ibuprofen 10 mg/kg orally (or through gastric tube) every 12 hours after surgery.
  In case of severe pain tramadol 0,5 mg/kg will be administered iv every 8 hours.

SUMMARY:
Effectiveness of the TAP block compared to wound infiltration in controlling pain after laparoscopic appendectomy in children

DETAILED DESCRIPTION:
Laparoscopic appendectomy is one of the main emergency surgical procedures performed in children.

The available local anesthesia techniques include wound infiltration or "wall" blocks such as the TAP (transversus abdominis plane) block.

The greater evidence on the adult population suggests that both techniques are valid for pain control in the immediate postoperative period, although wall blocks can guarantee a more prolonged analgesic effect over time.

The evidence on the pediatric population, on the other hand, is less strong and sometimes conflicting: therefore, the objective of our study is to verify the efficacy of TAP block compared to wound infiltration in the control of postoperative pain after appendectomy in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 3 and 16 years, candidates for laparoscopic appendectomy for suspected acute appendicitis.
* ASA physical status Class I and II
* Informed consent signed by parents / legal guardians

Exclusion Criteria:

* severe obesity (BMI> 95th percentile for age and weight)
* perforated appendicitis
* paralytic ileum
* non-stabilized neuropathies
* allergy to local anesthetics or analgesics used in the study protocol.
* patients on chronic opiate treatment
* need for perioperative hospitalization in intensive care with sedation and / or mechanical ventilation

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-03-30 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain at 2 hours | 2 hours
  Difference in pain severity (assessed by Wong Baker for under 8 year and visual analog scale dor older than 8) of TAP block goup compared to wound infiltration group 2 hours after the end of the surgery.

SECONDARY OUTCOMES:
Postoperative pain at 4-12-24 hours | from 4 to 24 postoperative hours
  Difference in pain severity (assessed by Wong Baker for under 8 year and visual analog scale dor older than 8) of TAP block goup compared to wound infiltration group 4 hours, 12 hours and 24 hours from the end of the surgery.
Total opioid consumption | from 2 to 24 postoperative hours
  Differences in tramadol rescue use (expressed in mg/kg) in the TAP group compared to the LIA group
time to first opioid analgesic rescue | from 2 to 24 postoperative hours
  Differences in the elapsed time before first request for tramadol rescue in the TAP group compared to the LIA group
Side effects | from 2 to 24 postoperative hours
  Differences in the incidence of side effects depending on the anesthetic technique adopted

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Day Surgery Ospedale di Circolo Varese, Varese, VA, Italy